CLINICAL TRIAL: NCT06606548
Title: The Impact of Comprehensive Oral Care on the Eating Function in Long-term Care Facilities Residents
Brief Title: Comprehensive Oral Care Long-term Care Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202305043RINC
Record Dates: First submitted 2024-06-13; First posted 2024-09-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dysphagia
Keywords: dysphagia; oral care; nasogastric tube
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general oral hygiene (No Intervention)
- comprehensive oral care (Experimental): including cleaning, facial massage, oral muscle massage and stretching, and oral moisturizing.
  Interventions: Behavioral: comprehensive oral care

INTERVENTIONS:
Behavioral: comprehensive oral care — including cleaning, facial massage, oral muscle massage and stretching, and oral moisturizing.
  Arms: comprehensive oral care

SUMMARY:
Oral care is a common way of caring for long-term care facility residents, particularly for those with swallowing difficulties, as oral health is closely related to eating function. Oral care includes general oral hygiene and comprehensive oral care (including cleaning, facial massage, oral muscle massage and stretching, and oral moisturizing). Regular oral care can reduce oral diseases, improve oral mucosa, increase appetite, and improve eating function. However, it is still unclear whether comprehensive oral care can improve eating function and aid in removing nasogastric tubes. Therefore, this study plans to recruit residents with dysphagia from multiple long-term care facilities nationwide to investigate the impact of comprehensive oral care on nasogastric tube removal. The study will collect basic information, disease diagnosis, and onset time and use random grouping to investigate the effects of general oral hygiene and oral care on nasogastric tube removal. The results of this study can provide guidance for clinical practitioners and researchers on oral care and eating function improvement for long-term care facility residents.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, with swallowing disorders classified as grades 1-3 on the Functional Oral Intake Scale (FOIS).
* Conscious and alert.
* Able to follow simple one-step commands (e.g., raising a hand, opening the mouth).
* Able to maintain a seated position for more than 15 minutes.
* Has a swallowing reflex (able to swallow saliva on command).

Exclusion Criteria:

* Acute infection.
* Hypoxemia (SaO2 < 90%) or requiring the use of a ventilator.
* Structural abnormalities of the oropharyngeal area that prevent oral feeding.
* Failing the water swallow test (coughing or wet voice in two or more out of three attempts, or no significant laryngeal elevation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Removing nasogastric tubes | Follow up for 6 months
  Each subject was tracked at one month, three months, and six months for the status of their nasogastric tube.

SECONDARY OUTCOMES:
the functional oral intake scale | Follow up for 6 months
body weight | Follow up for 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yen Hsiao, PHD, Principal Investigator — +886-2312-3456
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist., Taiwan

REFERENCES:
- [Result] Porter J, Ntouva A, Read A, Murdoch M, Ola D, Tsakos G. The impact of oral health on the quality of life of nursing home residents. Health Qual Life Outcomes. 2015 Jul 15;13:102. doi: 10.1186/s12955-015-0300-y. PMID 26169066
- [Result] Kenny A, Dickson-Swift V, Chan CKY, Masood M, Gussy M, Christian B, Hodge B, Furness S, Hanson LC, Clune S, Zadow E, Knevel RJ. Oral health interventions for older people in residential aged care facilities: a protocol for a realist systematic review. BMJ Open. 2021 May 5;11(5):e042937. doi: 10.1136/bmjopen-2020-042937. PMID 33952539
- [Result] Barbe AG, Kupeli LS, Hamacher S, Noack MJ. Impact of regular professional toothbrushing on oral health, related quality of life, and nutritional and cognitive status in nursing home residents. Int J Dent Hyg. 2020 Aug;18(3):238-250. doi: 10.1111/idh.12439. Epub 2020 May 11. PMID 32329175